CLINICAL TRIAL: NCT02052648
Title: A Phase I/II Study of the Combination of Indoximod and Temozolomide for Adult Patients With Temozolomide-Refractory Primary Malignant Brain Tumors
Brief Title: Study of IDO Inhibitor and Temozolomide for Adult Patients With Primary Malignant Brain Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NewLink Genetics Corporation (Industry)
Responsible Party: Sponsor
Organization: Lumos Pharma (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NLG2102
Record Dates: First submitted 2014-01-29; First posted 2014-02-03 (Estimated); Results first posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-02

CONDITIONS: Glioblastoma Multiforme; Glioma; Gliosarcoma; Malignant Brain Tumor
Keywords: glioblastoma multiforme; glioma; gliosarcoma; malignant brain tumor
MeSH Terms: conditions — Glioblastoma; Glioma; Gliosarcoma; Brain Neoplasms | interventions — 1-methyltryptophan; Temozolomide; Bevacizumab; Radiosurgery; Spermine Synthase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Phase 1b Cohort 1 (Experimental): Phase 1B patients will receive Indoximod given in escalating doses. Initial dosing will be 600 mg BID by mouth with escalation planned to 1200 mg BID by mouth. The medication should be taken twice daily for 28 days each cycle.
  Temozolomide will also be given by mouth at 150 mg/m^2 x 5 days at all dosing levels of indoximod. Each cycle is 28 days. Patients will continue until they experience disease progression or toxicity.
  Interventions: Drug: Indoximod; Drug: Temozolomide
- Cohort 2a (Experimental): Bevacizumab naïve phase II patients who will receive indoximod with temozolomide. Indoximod will be dosed at 1200mg BID. Temozolomide will be dosed at 150 mg/m2 and may be escalated up to 200 mg/m2.
  Interventions: Drug: Indoximod; Drug: Temozolomide
- Cohort 2b (Experimental): Phase II patients who will receive indoximod with temozolomide and bevacizumab who have previously been treated with bevacizumab.
  Indoximod will be dosed at 1200mg BID. Temozolomide will be dosed at 150 mg/m2 and may be escalated up to 200 mg/m2. Bevacizumab will be dosed at 10mg/kg.
  Interventions: Drug: Indoximod; Drug: Temozolomide; Drug: Bevacizumab
- Cohort 2c (Experimental): Phase II patients who will receive indoximod with temozolomide and stereotactic radiosurgery. Indoximod will be dosed at 1200mg BID. Temozolomide will be dosed at 150 mg/m2 and may be escalated up to 200 mg/m2. Single fraction SRS dose will be 16 or 20 Gy depending on target volume. The total 5-fraction SRT dose will be 27.5 Gy.
  Interventions: Drug: Indoximod; Drug: Temozolomide; Radiation: Stereotactic Radiation

INTERVENTIONS:
Drug: Indoximod
  Other Names: 1-methyl-D-tryptophan; D-1MT
Drug: Temozolomide
  Other Names: Temodar; Methazolastone
Drug: Bevacizumab
  Other Names: Avastin
  Arms: Cohort 2b
Radiation: Stereotactic Radiation
  Other Names: SRS or SRT
  Arms: Cohort 2c

SUMMARY:
In this study, investigators will conduct a phase I/II trial in recurrent (temozolomide resistant) glioma patients. The overall goal of this study is to provide a foundation for future studies with indoximod tested in newly diagnosed glioblastoma patients with radiation and temozolomide, or in combination with vaccine therapies.

DETAILED DESCRIPTION:
The aim of this study is to identify the safety profile and the recommended dose for phase 2 study of the combination of indoximod (portion 1, phase 1b study). Investigators will then evaluate the tolerability and the preliminary activity in patients with recurrent GBM in three different situations:

* Combination of indoximod and temozolomide (bevacizumab-naive patients)
* Combination of indoximod and temozolomide in patients currently receiving or having received and failed bevacizumab.
* Combination of indoximod and temozolomide with stereotactic radiation. Ancillary studies will be conducted to assess the correlation between intra-tumoral IDO expression or serum biomarkers (immune monitoring) and treatment efficacy.

If the current study shows an acceptable safety profile and suggests preliminary evidence of activity, this will provide the justification for subsequent randomized phase 2 studies in refractory glioblastoma multiforme (GBM).

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven intracranial glioblastoma multiforme (WHO grade IV glioma) or gliosarcoma. In addition, the Phase 1b cohort will include patients with progressive WHO grade III glioma.
* Patients will be eligible if the original histology was lower grade glioma and a subsequent diagnosis of glioblastoma or gliosarcoma is made.
* Unequivocal radiographic evidence for tumor progression by MRI. It is understood that some patients may be resected prior to enrolling onto protocol
* Patients must have completed a course of radiation therapy and at least 2 adjuvant cycles of temozolomide for the phase 2 component.
* Patients enrolling onto Cohort 2b who have been taken off bevacizumab must have had at least a 28 day washout from any previous administration of bevacizumab. It is preferred that patients who fail bevacizumab prior to trial entry remain on bevacizumab in the trial.
* Prior temozolomide is not required for the phase 1 component; prior radiation is required for the phase 1 arm.
* Patients must be on a steroid dose less than or equal to 2 mg of dexamethasone daily (or equivalent), and this dose must not have increased for at least 14 days prior to obtaining the enrollment.
* ECOG performance status ≤1 or Karnofsky ≥70%.
* Age between 16
* Must be 28 days from the administration of any investigational agent or prior cytotoxic therapy with the following exceptions:
* Must be 14 days from administration of non-cytotoxic agents (e.g., bevacizumab (except COHORT 2b), interferon, tamoxifen, thalidomide, cis-retinoic acid, tyrosine kinase inhibitor, etc.).

Exclusion Criteria:

* Prior invasive malignancy that is not low-grade glioma, high-grade glioma, glioblastoma, or gliosarcoma (except non-melanomatous skin cancer or carcinoma in situ of the cervix) unless the patient has been disease free and off therapy for that disease for a minimum of 3 years.
* Patients on the phase 2 portion of the study may not have more than 2 prior regimens for recurrent disease for glioblastoma/gliosarcoma. Patients on the phase 1 portion of the study may not have had more than 3 prior regimens.
* Systemic corticosteroid therapy > 2 mg of dexamethasone daily (or equivalent) at study enrollment.
* Active or history of autoimmune disease

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2014-03; Primary Completion 2018-04-18 (Actual); Study Completion 2019-06-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Eden Medical Center, Castro Valley, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - UC Irvine Chao Family Comprehensive Cancer Center, Orange, California
  - Moffitt Cancer Center, Tampa, Florida
  - University Cancer and Blood Center, Athens, Georgia
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Augusta University, Augusta, Georgia
  - University of Chicago, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kentucy, Lexington, Kentucky
  - John Nasseff Neuroscience Institute, Minneapolis, Minnesota
  - University of New Mexico Comprehensive Cancer Center, Albuquerque, New Mexico
  - Wake Forest Baptist Health Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Texas Oncology, Austin, Texas
  - Huntsman Cancer Center, Salt Lake City, Utah
  - Virginia Cancer Specialists, Fairfax, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1 Dose Level 1: Phase 1 Cohort 1 patients will receive Indoximod given at 600 mg BID by mouth Temozolomide will also be given by mouth at 150 mg/m^2 x 5 days
- Phase 1 Dose Level 2: Phase 1 Cohort 1 patients will receive Indoximod given at 1000 mg BID by mouth Temozolomide will also be given by mouth at 150 mg/m^2 x 5 days
- Phase 1 Dose Level 3: Phase 1 Cohort 1 patients will receive Indoximod given at 1200 mg BID by mouth Temozolomide will also be given by mouth at 150 mg/m^2 x 5 days
- Phase 2 Cohort 2a: Bevacizumab naïve phase II patients who will receive indoximod with temozolomide. Indoximod will be dosed at 1200mg BID. Temozolomide will be dosed at 150 mg/m2 and may be escalated up to 200 mg/m2.
- Phase 2 Cohort 2b: Phase II patients who will receive indoximod with temozolomide and bevacizumab who have previously been treated with bevacizumab.
  Indoximod will be dosed at 1200mg BID. Temozolomide will be dosed at 150 mg/m2 and may be escalated up to 200 mg/m2. Bevacizumab will be dosed at 10mg/kg.
- Phase 2 Cohort 2c: Phase II patients who will receive indoximod with temozolomide and stereotactic radiosurgery. Indoximod will be dosed at 1200mg BID. Temozolomide will be dosed at 150 mg/m2 and may be escalated up to 200 mg/m2. Single fraction SRS dose will be 16 or 20 Gy depending on target volume. The total 5-fraction SRT dose will be 27.5 Gy.
Period: Overall Study
Arm/Group | Phase 1 Dose Level 1 | Phase 1 Dose Level 2 | Phase 1 Dose Level 3 | Phase 2 Cohort 2a | Phase 2 Cohort 2b | Phase 2 Cohort 2c
Started | 3 | 3 | 6 | 80 | 28 | 40
Completed | 3 | 3 | 6 | 80 | 28 | 40
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1 Dose Level 1 | Phase 1 Dose Level 2 | Phase 1 Dose Level 3 | Phase 2 Cohort 2a | Phase 2 Cohort 2b | Phase 2 Cohort 2c | Total
Number analyzed (Participants) | 3 | 3 | 6 | 80 | 28 | 40 | 160
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 1 | 8 | 3 | 3 | 15
  Between 18 and 65 years | 3 | 3 | 5 | 53 | 17 | 31 | 112
  >=65 years | 0 | 0 | 0 | 19 | 8 | 6 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.7 (4.04) | 52.3 (12.66) | 48.0 (11.14) | 56.0 (13.69) | 54.0 (14.64) | 56.8 (12.20) | 55.2 (13.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 3 | 28 | 18 | 17 | 68
  Male | 1 | 3 | 3 | 52 | 10 | 23 | 92
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 8 | 1 | 1 | 10
  Not Hispanic or Latino | 3 | 3 | 5 | 68 | 27 | 39 | 145
  Unknown or Not Reported | 0 | 0 | 1 | 4 | 0 | 0 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 0 | 1 | 0 | 0 | 4
  White | 1 | 2 | 5 | 76 | 27 | 38 | 149
  More than one race | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 1 | 2 | 0 | 0 | 3
ECOG Performance Status Scale [Count of Participants; unit: Participants] — ECOG PERFORMANCE STATUS. Lower grade = better outcome.
  GRADE:
  0 = Fully active, able to carry on all pre-disease performance without restriction
  1. = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature
  2. = Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  3. = Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  4. = Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  5. = Dead
  Participants
    ECOG = 0 | 0 | 0 | 3 | 38 | 7 | 22 | 70
    ECOG = 1 | 3 | 2 | 3 | 37 | 20 | 17 | 82
    Missing | 0 | 1 | 0 | 5 | 1 | 1 | 8
Mean Height [Mean (Standard Deviation); unit: Centimeters] | 176.667 (12.6623) | 179.133 (5.5185) | 171.720 (8.8797) | 172.505 (9.8244) | 168.710 (9.3381) | 173.659 (10.1278) | 172.302 (9.839)
Mean Weight [Mean (Standard Deviation); unit: Kilograms] | 96.467 (22.7315) | 103.117 (22.9877) | 81.083 (25.0460) | 83.342 (17.5121) | 75.882 (11.5149) | 84.649 (19.2743) | 82.895 (17.881)
Mean BMI [Mean (Standard Deviation); unit: kg/m2] | 31.807 (11.9796) | 31.967 (5.1495) | 27.260 (7.894) | 27.904 (5.1508) | 26.633 (3.5701) | 28.037 (6.0775) | 27.84 (5.42)

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Regimen-Limiting Toxicities (RLTs) in Phase 1 Subjects
Description: Number of RLTs observed in each dose level.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Dose Level 1 | Phase 1 Dose Level 2 | Phase 1 Dose Level 3
Number analyzed (Participants) | 3 | 3 | 6
Participants | 0 | 0 | 0

2. Primary Outcome: Phase 2: Number of Phase 1 Participants With Efficacy Outcomes
Description: Six-month progression-free survival.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: Percent
Arm/Group | Phase 2 Cohort 2a | Phase 2 Cohort 2b | Phase 2 Cohort 2c
Number analyzed (Participants) | 77 | 28 | 39
Percent | 18.6 [10.4 to 28.8] | 3.9 [0.3 to 16.6] | 22.9 [10.5 to 38.3]

3. Secondary Outcome: Overall Response Rate for Phase 2 Participants
Description: Subjects with a complete response or partial response by RANO assessment. Overall Response Rate was only assessed in phase 2 subjects on this trial.
Time Frame: 18 months
Measure: Number (95% Confidence Interval); unit: Percent
Arm/Group | Phase 2 Cohort 2a | Phase 2 Cohort 2b | Phase 2 Cohort 2c
Number analyzed (Participants) | 77 | 28 | 39
Percent | 5.2 [1.4 to 12.8] | 0 [0 to 12.3] | 7.7 [1.6 to 20.9]

4. Secondary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Description: Number of subjects with at least 1 treatment emergent adverse event.
Time Frame: 18 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Dose Level 1 | Phase 1 Dose Level 2 | Phase 1 Dose Level 3 | Phase 2 Cohort 2a | Phase 2 Cohort 2b | Phase 2 Cohort 2c
Number analyzed (Participants) | 3 | 3 | 6 | 77 | 28 | 39
Participants | 3 | 3 | 6 | 72 | 27 | 39

ADVERSE EVENTS:
Time Frame: Up to 36 months.
Arm/Group | Phase 1 Dose Level 1 | Phase 1 Dose Level 2 | Phase 1 Dose Level 3 | Phase 2 Cohort 2a | Phase 2 Cohort 2b | Phase 2 Cohort 2c
All-Cause Mortality (participants affected / at risk) | 3/3 | 3/3 | 6/6 | 67/77 | 28/28 | 34/39
Serious Adverse Events (participants affected / at risk) | 2/3 | 1/3 | 1/6 | 21/77 | 10/28 | 17/39
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 6/6 | 77/77 | 28/28 | 39/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Dose Level 1 (N=3) | Phase 1 Dose Level 2 (N=3) | Phase 1 Dose Level 3 (N=6) | Phase 2 Cohort 2a (N=77) | Phase 2 Cohort 2b (N=28) | Phase 2 Cohort 2c (N=39)
Seizure (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 6 (6)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 4 (4)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Partial seizures (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Radiation necrosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Dose Level 1 (N=3) | Phase 1 Dose Level 2 (N=3) | Phase 1 Dose Level 3 (N=6) | Phase 2 Cohort 2a (N=77) | Phase 2 Cohort 2b (N=28) | Phase 2 Cohort 2c (N=39)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 4 (4) | 22 (22) | 7 (7) | 19 (19)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2) | 13 (13) | 1 (1) | 5 (5)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 12 (12) | 3 (3) | 8 (8)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 10 (10) | 5 (5) | 9 (9)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 9 (9) | 1 (1) | 4 (4)
Seizure (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 9 (9) | 2 (2) | 12 (12)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 6 (6) | 2 (2) | 7 (7)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 4 (4)
Visual field defect (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Neurologic neglect syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Aura (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Clonus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diplegia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyscalculia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyskinesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dysmetria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 | 0 | 2
Facial paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 3 (3)
Facial paresis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hemianopia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemianopia homonymous (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypersomnia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post herpetic neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Psychomotor skills impaired (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper motor neurone lesion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Apraxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Drooling (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Head discomfort (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperreflexia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Partial seizures (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Postictal paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sensory loss (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tardive dyskinesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 | 3 | 4 | 54 | 19 | 21
Constipation (Gastrointestinal disorders) | 2 | 1 | 0 | 34 (34) | 7 (7) | 20 (20)
Vomiting (Gastrointestinal disorders) | 1 | 3 | 4 | 25 (25) | 8 (8) | 14 (14)
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 8 (8) | 4 (4) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 3 (3) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 6 (6)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proctitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 | 0 | 0
Colitis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lip swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Glossitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral dysaesthesia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 2 (2) | 31 (31) | 9 (9) | 21 (21)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 1 (1) | 4 (4) | 4 (4) | 2 (2)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 3 (3) | 3 (3)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 11 (11) | 1 (1) | 5 (5)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 7 (7) | 1 (1) | 5 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 4 (4) | 2 (2) | 1 (1)
Hyperchloraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 9 (9) | 4 (4) | 5 (5)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 3 (3) | 2 (2)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 8 (8) | 4 (4) | 11 (11)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 2 (2)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 5 (5) | 2 (2) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 0 (0) | 3 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 3 (3)
Bone lesion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Posture abnormal (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1) | 5 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 6 (6)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 6 (6)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary necrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 6 (6) | 1 (1) | 3 (3)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Photopsia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythema of eyelid (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ocular discomfort (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 7 (7) | 2 (2) | 9 (9)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 2 (2) | 4 (4)
Personality change (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 1 (1) | 4 (4)
Abulia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Affect lability (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Frustration tolerance (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Phonophobia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bruxism (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1
Hallucination,Visual (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1
Mania (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 9 (9) | 5 (5) | 8 (8)
Mood altered (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 0 (0) | 3 (3)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Angular cheilitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Escherichia infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nail infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 2 (2) | 8 (8)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 7 (7)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Precancerous skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 3 (3)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 4 (4)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural persistent drain fluid (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Incision site pain s (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural anxiety (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 18 (18) | 7 (7) | 9 (9)
Skin abrasion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Radiation necrosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tongue injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 5 (5) | 4 (4) | 3 (3)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chromaturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Motion sickness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Deafness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (12)
Inner ear disorder (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Middle ear effusion (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Bundle branch block right (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Cushingoid (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Scrotal oedema (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 8 (8) | 3 (3) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 0 (0) | 5 (5)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 13 (13) | 4 (4) | 4 (4)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 1 (1) | 4 (4)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 1 (1) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 4 (4)
Alanine aminotransferase increase (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased blood (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood potassium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prothrombin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood chloride decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Head lag abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2015-08-27): https://cdn.clinicaltrials.gov/large-docs/48/NCT02052648/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-18): https://cdn.clinicaltrials.gov/large-docs/48/NCT02052648/SAP_001.pdf